CLINICAL TRIAL: NCT00818961
Title: Reduced Intensity Allogeneic Stem Cell Transplantation With Matched Unrelated Donors for Patients With Hematologic Malignancies
Brief Title: Donor Stem Cell Transplant in Treating Patients With High-Risk Hematologic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: terminated early due to meeting end point with fewer patients than anticipated
Sponsor: Northside Hospital, Inc. (Other)
Collaborators: Blood and Marrow Transplant Group of Georgia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000630617; BMTGG-NSH-756 (Other: Northside Hospital, Inc)
Record Dates: First submitted 2009-01-07; First posted 2009-01-08 (Estimated); Results first posted 2013-12-18 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-10

CONDITIONS: Leukemia; Lymphoma; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases
Keywords: accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; adult AML with 11q23 (MLL) abnormalities; blastic phase chronic myelogenous leukemia; chronic myelomonocytic leukemia; chronic phase chronic myelogenous leukemia; prolymphocytic leukemia; recurrent adult T-cell leukemia/lymphoma; refractory chronic lymphocytic leukemia; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; stage I adult T-cell leukemia/lymphoma; stage I chronic lymphocytic leukemia; stage II adult T-cell leukemia/lymphoma; stage II chronic lymphocytic leukemia; stage III adult T-cell leukemia/lymphoma; stage III chronic lymphocytic leukemia; stage IV adult T-cell leukemia/lymphoma; stage IV chronic lymphocytic leukemia; recurrent adult Hodgkin lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; cutaneous B-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell NHL; stage I cutaneous T-cell NHL; stage II cutaneous T-cell NHL; stage III cutaneous T-cell NHL; stage IV cutaneous T-cell NHL; extranodal marginal zone B-cell lymphoma of mucosal tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; contiguous st II adult diffuse large cell lymphoma; contiguous st II adult diffuse mixed cell lymphoma; contiguous st II adult diffuse sm cleaved cell lymphoma; contiguous st II grade 1 follicular lymphoma; contiguous st II grade 2 follicular lymphoma; contiguous st II grade 3 follicular lymphoma; contiguous st II mantle cell lymphoma; contiguous st II marginal zone lymphoma; contiguous st II small lymphocytic lymphoma; stage I adult diffuse large cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I mantle cell lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; noncontiguous st II adult diffuse large cell lymphoma; noncontiguous st II adult diffuse mixed cell lymphoma; noncontiguous st II adult diffuse sm cleaved cell lymphoma; noncontiguous st II grade 1 follicular lymphoma; noncontiguous st II grade 2 follicular lymphoma; noncontiguous st II grade 3 follicular lymphoma; noncontiguous st II mantle cell lymphoma; noncontiguous st II marginal zone lymphoma; noncontiguous st II small lymphocytic lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult gr III lymphomatoid granulomatosis; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; de novo MDS; previously treated MDS; secondary myelodysplastic syndromes; Waldenstrom macroglobulinemia; myelodysplastic/myeloproliferative disease
MeSH Terms: conditions — Leukemia; Lymphoma; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Prolymphocytic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Hodgkin Disease; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Waldenstrom Macroglobulinemia | interventions — Alemtuzumab; Rituximab; Busulfan; Cyclophosphamide; fludarabine phosphate; Methotrexate; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hematopoietic Stem Cell Transplantation (Other): All patients receive a hematopoietic stem cell transplant using one of two chemotherapy regimens based on donor type
  Interventions: Biological: alemtuzumab; Biological: graft-versus-tumor induction therapy; Biological: rituximab; Drug: busulfan; Drug: cyclophosphamide; Drug: fludarabine phosphate; Drug: methotrexate; Drug: tacrolimus; Procedure: allogeneic bone marrow transplantation

INTERVENTIONS:
Biological: alemtuzumab — 43 mg subcutaneously over 3 days (3 mg on day -11, 10 mg on day -10, 30 mg on day -9)
  Other Names: Campath
Biological: graft-versus-tumor induction therapy — curative potential of allogeneic transplant results from the immune anti-tumor effect of donor cells or GVT/GVL
Biological: rituximab — in patients with Cd20+ malignancies: rituximab 375 mg/m*2 day -13. rituximab 1000 mg/m*2 on days, -6, +1, +8.
  Other Names: Rituxan
Drug: busulfan — For patients with AML, CML, MDS, MPS and ALL only: IV or oral busulfan may be given IV busulfan: 130 mg/m2 over 3 hours once daily on days -6, -5, -4 and -3 Oral busulfan: taken every 6 hours x 15 doses beginning on day -7 at 6pm and continuing through day -3 at 6am. 1 mg/kg test dose will be given prior to day -7 and PK samples will be drawn to calculate AUC.
Drug: cyclophosphamide — 750 mg/m2 infused over 1 hour once daily on days -5, -4 and -3. Cyclophosphamide will be started approximately 4 hours after the start of Fludarabine
  Other Names: Cytoxan
Drug: fludarabine phosphate — For patients with CLL, NHL & HD: 30 mg/m2 infused over 30 minutes once daily on days -5, -4 and -3 For patients with AML, CML, MDS, MPS and ALL: 40 mg/m2 infused over 30 minutes once daily on days -6, -5, -4 and -3.
  Other Names: Fludara
Drug: methotrexate — 5 mg/m2 administered on days +1, +3 and +6
Drug: tacrolimus — 0.03mg/kg/day infused over 24 hours starting on day -1 and switched to oral (twice daily divided dose) on day 14 or when able to tolerate PO
  Other Names: Prograf; FK506
Procedure: allogeneic bone marrow transplantation — Recipients will receive an allogeneic transplant on day 0 after receiving high-dose chemotherapy. This trial uses matched unrelated donor stem cells.
  Other Names: HSCT, allo transplant

SUMMARY:
RATIONALE: Giving low doses of chemotherapy before a donor stem cell transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving a monoclonal antibody, such as alemtuzumab, before transplant and tacrolimus and methotrexate after transplant may stop this from happening.

PURPOSE: This phase II trial is studying the side effects of donor stem cell transplant and to see how well it works in treating patients with high-risk hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the safety and toxicity of a reduced-intensity conditioning regimen followed by allogeneic bone marrow or peripheral blood stem cell transplantation from an HLA-matched unrelated donor in patients with high-risk hematologic malignancies.
* To evaluate engraftment by peripheral blood chimerism analysis.
* To determine the incidence and severity of acute and chronic graft-versus-host disease following the transplant.
* To examine the possibility of controlling hematologic malignancies by induction of a graft-versus-leukemia/tumor effect.
* To determine the disease-free survival, relapse, transplant-related mortality, and death from all causes.

OUTLINE:

* Reduced-intensity conditioning regimen: Patients receive 1 of 2 conditioning regimens according to diagnosis.

  * Regimen 1 (acute leukemia, myelodysplastic syndromes, myeloproliferative syndrome, or chronic myelogenous leukemia): Patients receive fludarabine phosphate IV over 30 minutes and busulfan IV over 3 hours on days -6 to -3 or orally 4 times daily on days -7 to -3.
  * Regimen 2 (lymphoproliferative malignancies): Patients receive fludarabine phosphate IV over 30 minutes and cyclophosphamide IV over 1 hour on days -5 to -3. Patients with CD20+ malignancies also receive rituximab IV over 4-6 hours on days -13, -6, 1, and 8.
* Transplantation: Patients undergo allogeneic bone marrow or peripheral blood stem cell transplantation on day 0.
* Graft-versus-host disease (GVHD) prophylaxis: Patients receive low-dose alemtuzumab subcutaneously on days -11 to -9 and tacrolimus IV over 24 hours beginning on day -3 and then orally twice daily beginning on day 14 and continuing until day 60, followed by a taper until day 180 in the absence of clinically significant GVHD. Patients also receive methotrexate on days 1, 3, and 6.

Patients who exhibit persistent mixed chimerism or disease relapse/progression despite full withdrawal of immunosuppression may receive up to 3 donor lymphocyte infusions.

Blood samples are taken on days 30, 60, and 100 and then every 4 weeks thereafter for chimerism studies by PCR analysis.

After completion of study therapy, patients are followed periodically for up to 60 months.

ELIGIBILITY:
* Diagnosis of one of the following hematological malignancies:

  * CML, with 1 of the following:

    * In first CP AND failed imatinib mesylate therapy, defined as failure to obtain a hematologic remission at 3 months or a major cytogenetic response (i.e., Ph+ cells < 35%) at 6 months or demonstrated clonal evolution or disease progression during therapy
    * In accelerated phase with < 15% blasts
    * In blast crisis that has entered into a second CP following induction chemotherapy
  * AML, with 1 of the following:

    * In second or subsequent complete remission (CR) (i.e., < 5% blasts by morphology, no residual leukemia by flow cytometry, and absence of cytogenetic abnormalities)
    * Failed primary induction chemotherapy, but subsequently entered into a CR with ≤ 2 subsequent re-induction chemotherapy treatment(s)
    * In first CR with intermediate-risk or poor-risk cytogenetics
  * ALL with 1 of the following:

    * In second or subsequent CR
    * In first CR AND presence of t(9;22)
  * MDS, with the following:

    * High-risk disease, defined by IPSS score of ≥ 1.5 at diagnosis AND meets 1 of the following criteria:

      * ≤ 10% blasts at diagnosis
      * In morphologic CR (< 5% blasts) following cytoreductive chemotherapy
  * CMML, with 1 of the following:

    * ≤ 10% blasts at diagnosis
    * In morphologic CR (< 5% blasts) following cytoreductive chemotherapy
  * CLL/PLL with the following:

    * Rai stage I-IV disease
    * Failed ≥ 1 prior chemotherapy regimen (including fludarabine phosphate) or ASCT
    * Documented chemosensitive or stable, non-bulky disease prior to transplant, defined as < 20% bone marrow involvement AND lymph node size < 3 cm in axial diameter
    * No bulky tumor masses, elevated lactate dehydrogenase (LDH), B symptoms, or progressive disease prior to transplant
  * Low-grade non-Hodgkin lymphoma (NHL) (i.e., small lymphocytic lymphoma, follicular center lymphoma [grade 1 or 2], marginal zone lymphoma, or B-cell lymphoma), with the following criteria:

    * Failed ≥ 1 prior chemotherapy regimen or ASCT
    * Documented chemosensitive or stable, non-bulky disease prior to transplant, defined as < 20% bone marrow involvement AND lymph node size < 3 cm in axial diameter
    * Received ≤ 3 prior chemotherapy regimens (monoclonal antibody therapy and involved-field radiotherapy are not considered a prior regimen)
    * No bulky tumor masses, elevated LDH, B symptoms, or progressive disease prior to transplant
  * Mantle cell lymphoma, with the following:

    * Failed to achieve remission or recurred after either conventional chemotherapy or ASCT
    * Responsive or stable disease to most recent prior therapy
    * No bulky tumor masses, elevated LDH, B symptoms, or progressive disease prior to transplant
  * Intermediate-grade NHL (i.e., follicular center lymphoma [grade 3] or diffuse large cell lymphoma), meeting the following criteria:

    * Failed to achieve remission or recurred after either conventional chemotherapy or ASCT
    * Documented chemosensitive, non-bulky disease prior to transplant, defined as at least a partial remission to salvage chemotherapy (≥ 50% reduction in diameter of all disease sites)
    * No bulky tumor masses, elevated LDH, B symptoms, or progressive disease prior to transplant
  * Hodgkin lymphoma, with the following:

    * Relapsed after prior ASCT OR after ≥ 2 combination chemotherapy regimens and ineligible for ASCT
    * Documented chemosensitive, non-bulky disease prior to transplant, defined as at least a partial remission to salvage chemotherapy (≥ 50% reduction in diameter of all disease sites)
    * No bulky tumor masses, elevated LDH, B symptoms, or progressive disease prior to transplant
  * Peripheral T-cell NHL, with the following:

    * Failed to achieve remission or recurred after either conventional chemotherapy or ASCT
    * Documented chemosensitive, non-bulky disease prior to transplant, defined as at least a partial remission to salvage chemotherapy (≥ 50% reduction in diameter of all disease sites)
    * No bulky tumor masses, elevated LDH, B symptoms, or progressive disease prior to transplant
* Myeloproliferative syndrome with poor risk features, meeting 1 of the following criteria:

  * < 55 years old AND Lille score of 1
  * Lille score of 2
  * HgB < 10 g/dL AND abnormal karyotype
* High-risk disease, with 1 of the following:

  * Age 40-72 years
  * Any age AND deemed to be at significantly increased risk of morbidity and death following a standard, myeloablative unrelated donor stem cell transplant (e.g., received extensive prior therapy, including ASCT)
* HLA-matched unrelated donor available, with 1 of the following:

  * 8/8 match at HLA-A, B, C, or DR loci by high-resolution genotyping
  * Single allelic mismatch at either the HLA-B or HLA-C loci donor by high-resolution molecular typing

    * No single allelic mismatch at HLA-A or HLA-DR loci
* KPS 80-100%
* Adapted weighted Charlson Comorbidity Index < 3
* Serum creatinine ≤ 2.0 mg/dL
* AST or ALT < 3 times upper limit of normal (ULN)
* Total bilirubin < 1.5 times ULN
* LVEF ≥ 45%
* DLCO > 50%
* No hypoxia at rest with oxygen saturation < 92% on room air (corrected with bronchodilator therapy)
* No other severe pulmonary function abnormalities
* No HIV infection
* No active hepatitis B or C infection that, in the opinion of a gastroenterologist or the transplant committee, places the patient at moderate to high risk for developing severe hepatic disease
* No active opportunistic infection (e.g., fungal pneumonia, tuberculosis, or viral infection)

Ages: 40 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-05; Primary Completion 2011-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott R. Solomon, MD, Principal Investigator — Blood and Marrow Transplant Group of Georgia
Locations (1):
- Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia, United States

REFERENCES:
- [Background] McGlave PB, Shu XO, Wen W, Anasetti C, Nademanee A, Champlin R, Antin JH, Kernan NA, King R, Weisdorf DJ. Unrelated donor marrow transplantation for chronic myelogenous leukemia: 9 years' experience of the national marrow donor program. Blood. 2000 Apr 1;95(7):2219-25. PMID 10733488
- [Background] Sierra J, Storer B, Hansen JA, Martin PJ, Petersdorf EW, Woolfrey A, Matthews D, Sanders JE, Storb R, Appelbaum FR, Anasetti C. Unrelated donor marrow transplantation for acute myeloid leukemia: an update of the Seattle experience. Bone Marrow Transplant. 2000 Aug;26(4):397-404. doi: 10.1038/sj.bmt.1702519. PMID 10982286
- [Background] Weisdorf DJ, Billett AL, Hannan P, Ritz J, Sallan SE, Steinbuch M, Ramsay NK. Autologous versus unrelated donor allogeneic marrow transplantation for acute lymphoblastic leukemia. Blood. 1997 Oct 15;90(8):2962-8. PMID 9376576
- [Background] Anderson JE, Anasetti C, Appelbaum FR, Schoch G, Gooley TA, Hansen JA, Buckner CD, Sanders JE, Sullivan KM, Storb R. Unrelated donor marrow transplantation for myelodysplasia (MDS) and MDS-related acute myeloid leukaemia. Br J Haematol. 1996 Apr;93(1):59-67. doi: 10.1046/j.1365-2141.1996.4811022.x. PMID 8611476
- [Background] Izutsu K, Kanda Y, Ohno H, Sao H, Ogawa H, Miyazaki Y, Kawa K, Kodera Y, Kato S, Morishima Y, Hirai H; Japan Marrow Donor Program. Unrelated bone marrow transplantation for non-Hodgkin lymphoma: a study from the Japan Marrow Donor Program. Blood. 2004 Mar 1;103(5):1955-60. doi: 10.1182/blood-2003-03-0937. Epub 2003 Nov 6. PMID 14604976
- [Background] Shaw BE, Peggs K, Bird JM, Cavenagh J, Hunter A, Alejandro Madrigal J, Russell NH, Sirohi B, Towlson K, Williams CD, Marks DI; Clinical Trials Committee of the British Society of Blood and Marrow Transplantation. The outcome of unrelated donor stem cell transplantation for patients with multiple myeloma. Br J Haematol. 2003 Dec;123(5):886-95. doi: 10.1046/j.1365-2141.2003.04714.x. PMID 14632780
- [Background] Davies SM, Kollman C, Anasetti C, Antin JH, Gajewski J, Casper JT, Nademanee A, Noreen H, King R, Confer D, Kernan NA. Engraftment and survival after unrelated-donor bone marrow transplantation: a report from the national marrow donor program. Blood. 2000 Dec 15;96(13):4096-102. PMID 11110679
- [Background] Hansen JA, Gooley TA, Martin PJ, Appelbaum F, Chauncey TR, Clift RA, Petersdorf EW, Radich J, Sanders JE, Storb RF, Sullivan KM, Anasetti C. Bone marrow transplants from unrelated donors for patients with chronic myeloid leukemia. N Engl J Med. 1998 Apr 2;338(14):962-8. doi: 10.1056/NEJM199804023381405. PMID 9521984
- [Background] Sorror ML, Maris MB, Storer B, Sandmaier BM, Diaconescu R, Flowers C, Maloney DG, Storb R. Comparing morbidity and mortality of HLA-matched unrelated donor hematopoietic cell transplantation after nonmyeloablative and myeloablative conditioning: influence of pretransplantation comorbidities. Blood. 2004 Aug 15;104(4):961-8. doi: 10.1182/blood-2004-02-0545. Epub 2004 Apr 27. PMID 15113759
- [Background] Sullivan KM, Weiden PL, Storb R, Witherspoon RP, Fefer A, Fisher L, Buckner CD, Anasetti C, Appelbaum FR, Badger C, et al. Influence of acute and chronic graft-versus-host disease on relapse and survival after bone marrow transplantation from HLA-identical siblings as treatment of acute and chronic leukemia. Blood. 1989 May 1;73(6):1720-8. PMID 2653460
- [Background] Mehta J, Singhal S. Graft-versus-myeloma. Bone Marrow Transplant. 1998 Nov;22(9):835-43. doi: 10.1038/sj.bmt.1701459. PMID 9827810
- [Background] Jones RJ, Ambinder RF, Piantadosi S, Santos GW. Evidence of a graft-versus-lymphoma effect associated with allogeneic bone marrow transplantation. Blood. 1991 Feb 1;77(3):649-53. PMID 1991174
- [Background] Porter DL, Connors JM, Van Deerlin VM, Duffy KM, McGarigle C, Saidman SL, Leonard DG, Antin JH. Graft-versus-tumor induction with donor leukocyte infusions as primary therapy for patients with malignancies. J Clin Oncol. 1999 Apr;17(4):1234. doi: 10.1200/JCO.1999.17.4.1234. PMID 10561184
- [Background] O'Brien S, Kantarjian H, Beran M, Smith T, Koller C, Estey E, Robertson LE, Lerner S, Keating M. Results of fludarabine and prednisone therapy in 264 patients with chronic lymphocytic leukemia with multivariate analysis-derived prognostic model for response to treatment. Blood. 1993 Sep 15;82(6):1695-700. PMID 8400226
- [Background] Giralt S, Estey E, Albitar M, van Besien K, Rondon G, Anderlini P, O'Brien S, Khouri I, Gajewski J, Mehra R, Claxton D, Andersson B, Beran M, Przepiorka D, Koller C, Kornblau S, Korbling M, Keating M, Kantarjian H, Champlin R. Engraftment of allogeneic hematopoietic progenitor cells with purine analog-containing chemotherapy: harnessing graft-versus-leukemia without myeloablative therapy. Blood. 1997 Jun 15;89(12):4531-6. PMID 9192777
- [Background] Diaconescu R, Flowers CR, Storer B, Sorror ML, Maris MB, Maloney DG, Sandmaier BM, Storb R. Morbidity and mortality with nonmyeloablative compared with myeloablative conditioning before hematopoietic cell transplantation from HLA-matched related donors. Blood. 2004 Sep 1;104(5):1550-8. doi: 10.1182/blood-2004-03-0804. Epub 2004 May 18. PMID 15150081
- [Background] Escalon MP, Champlin RE, Saliba RM, Acholonu SA, Hosing C, Fayad L, Giralt S, Ueno NT, Maadani F, Pro B, Donato M, McLaughlin P, Khouri IF. Nonmyeloablative allogeneic hematopoietic transplantation: a promising salvage therapy for patients with non-Hodgkin's lymphoma whose disease has failed a prior autologous transplantation. J Clin Oncol. 2004 Jun 15;22(12):2419-23. doi: 10.1200/JCO.2004.09.092. PMID 15197204
- [Background] Khouri IF, Lee MS, Saliba RM, Andersson B, Anderlini P, Couriel D, Hosing C, Giralt S, Korbling M, McMannis J, Keating MJ, Champlin RE. Nonablative allogeneic stem cell transplantation for chronic lymphocytic leukemia: impact of rituximab on immunomodulation and survival. Exp Hematol. 2004 Jan;32(1):28-35. doi: 10.1016/j.exphem.2003.09.021. PMID 14725898
- [Background] Kernan NA, Bartsch G, Ash RC, Beatty PG, Champlin R, Filipovich A, Gajewski J, Hansen JA, Henslee-Downey J, McCullough J, et al. Analysis of 462 transplantations from unrelated donors facilitated by the National Marrow Donor Program. N Engl J Med. 1993 Mar 4;328(9):593-602. doi: 10.1056/NEJM199303043280901. PMID 8429851
- [Background] Champlin RE, Passweg JR, Zhang MJ, Rowlings PA, Pelz CJ, Atkinson KA, Barrett AJ, Cahn JY, Drobyski WR, Gale RP, Goldman JM, Gratwohl A, Gordon-Smith EC, Henslee-Downey PJ, Herzig RH, Klein JP, Marmont AM, O'Reilly RJ, Ringden O, Slavin S, Sobocinski KA, Speck B, Weiner RS, Horowitz MM. T-cell depletion of bone marrow transplants for leukemia from donors other than HLA-identical siblings: advantage of T-cell antibodies with narrow specificities. Blood. 2000 Jun 15;95(12):3996-4003. PMID 10845940
- [Background] Perez-Simon JA, Kottaridis PD, Martino R, Craddock C, Caballero D, Chopra R, Garcia-Conde J, Milligan DW, Schey S, Urbano-Ispizua A, Parker A, Leon A, Yong K, Sureda A, Hunter A, Sierra J, Goldstone AH, Linch DC, San Miguel JF, Mackinnon S; Spanish and United Kingdom Collaborative Groups for Nonmyeloablative Transplantation. Nonmyeloablative transplantation with or without alemtuzumab: comparison between 2 prospective studies in patients with lymphoproliferative disorders. Blood. 2002 Nov 1;100(9):3121-7. doi: 10.1182/blood-2002-03-0701. PMID 12384408
- [Background] Byrne JL, Stainer C, Cull G, Haynes AP, Bessell EM, Hale G, Waldmann H, Russell NH. The effect of the serotherapy regimen used and the marrow cell dose received on rejection, graft-versus-host disease and outcome following unrelated donor bone marrow transplantation for leukaemia. Bone Marrow Transplant. 2000 Feb;25(4):411-7. doi: 10.1038/sj.bmt.1702165. PMID 10723585
- [Background] Faulkner RD, Craddock C, Byrne JL, Mahendra P, Haynes AP, Prentice HG, Potter M, Pagliuca A, Ho A, Devereux S, McQuaker G, Mufti G, Yin JL, Russell NH. BEAM-alemtuzumab reduced-intensity allogeneic stem cell transplantation for lymphoproliferative diseases: GVHD, toxicity, and survival in 65 patients. Blood. 2004 Jan 15;103(2):428-34. doi: 10.1182/blood-2003-05-1406. Epub 2003 Sep 11. PMID 12969983

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient on this study was enrolled & transplanted on 6/9/05. The last patient on this study was enrolled & transplanted on 1/5/11.
Pre-assignment Details: No "groups" were assigned. Pts received chemotherapy based on their disease. 39 patients consented to study but 36 patients received protocol treatment. 3 patients were considered screen failures and did not move forward on study.
Groups:
- Hematopoietic Stem Cell Transplantation: All patients receive a hematopoietic stem cell transplant using one of two chemotherapy regimens based on disease type
Period: Overall Study
Arm/Group | Hematopoietic Stem Cell Transplantation
Started | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 56.44 (6.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Survival at Day 100
Description: Survival at Day 100
Time Frame: 100 day
Population: 36 patients underwent hematopoietic stem cell transplant and therefore were eligible for evaluation of overall survival at 100 days
Measure: Number; unit: participants
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 36
participants | 35

2. Secondary Outcome: Overall Survival at 1 Year
Description: Evaluation of overall survival at 1 year (# of patients who are alive at 1 year post-transplant)
Time Frame: 1 year
Population: 36 patients underwent hematopoietic stem cell transplant and therefore were eligible for evaluation of overall survival at one year post-transplant
Measure: Number; unit: participants
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 36
participants | 26

3. Secondary Outcome: Non-relapse Mortality at Day 100
Description: patients are evaluable for their cause of death at Day 100
Time Frame: Day 100
Population: 36 patients underwent hematopoietic stem cell transplant and therefore were eligible for evaluation of non-relapse mortality at Day 100
Measure: Number; unit: participants
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 36
participants | 1

4. Secondary Outcome: Non-relapse Mortality at 1 Year Post-transplant
Description: Number of patients who died of non-relapse causes at one year. this is in clusive of all patients who were transplanted on study even though only 10 patients died at by 1 year time point. This outcome will be referenced in the donor chimerism outcome. Only 26/36 patients were eligible for this time point as that is all that were alive.
Time Frame: 1 year
Population: 36 patients underwent hematopoietic stem cell transplant. 10 patients died prior to 1 year post-transplant and were eligible for evaluation of non-relapse mortality at 1 year post-transplant
Measure: Number; unit: participants
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 36
participants | 4

5. Secondary Outcome: Complete Donor Chimerism
Description: Complete donor chimerism (defined as >/= 95% donor cells in peripheral blood CD3+ and CD33+ was measured.
Time Frame: 2 years
Population: 36 patients underwent hematopoietic stem cell transplant and therefore were eligible for evaluation of donor chimerism
Measure: Number; unit: participants
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 36
participants | 26

6. Secondary Outcome: Neutrophil Recovery
Description: The number of patients experiencing neutrophil recovery post transplant
Time Frame: Day 100
Population: 36 patients underwent hematopoietic stem cell transplant and therefore were eligible for evaluation of neutrophil recovery
Measure: Number; unit: participants
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 36
participants | 35

7. Secondary Outcome: Platelet Engraftment
Description: The number of patients experiencing platelet engraftment post-transplant
Time Frame: Day 100
Population: 36 patients underwent hematopoietic stem cell transplant and therefore were eligible for evaluation of platelet engraftment.
Measure: Number; unit: participants
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 36
participants | 35

8. Secondary Outcome: Number of Patients Requiring the Use of Donor Leukocyte Infusion (DLI) for Early Mixed T-cell Chimerism
Description: DLI is used for patients with mixed chimerism following transplant
Time Frame: Day 100
Population: 36 patients underwent hematopoietic stem cell transplant and therefore were eligible for donor leukocyte infusions for mixed chimerism following transplant
Measure: Number; unit: participants
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 36
participants | 19

9. Secondary Outcome: Number of Patients Experiencing Grade 2-4 Acute Graft-versus-host Disease Post-transplant
Description: patients experiencing acute graft versus host disease post-transplant
Time Frame: patients were followed for 2 years
Population: 36 patients underwent hematopoietic stem cell transplant and therefore were eligible for evaluation of acute graft versus host disease post-transplant.
Measure: Number; unit: participants
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 36
participants | 15

10. Secondary Outcome: Number of Patients Experiencing Chronic Graft Versus Host Disease
Time Frame: >100 days post-transplant
Population: 35 patients survive past 100 days post-transplant and therefore were eligible for evaluation of chronic graft versus host disease
Measure: Number; unit: participants
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 35
participants | 20

11. Secondary Outcome: Number of Patients Experiencing Veno-occlusive Disease (VOD) Post-transplant
Description: Patients will be evaluated up to 4 years post transplant
Time Frame: 4 years
Population: 36 patients underwent hematopoietic stem cell transplant and therefore were eligible for evaluation of VOD post-transplant
Measure: Number; unit: participants
Arm/Group | Hematopoietic Stem Cell Transplantation
Number analyzed (Participants) | 36
participants | 0

ADVERSE EVENTS:
Groups:
- Hematopoietic Stem Cell Transplantation: All patients received a hematopoietic Stem Cell Transplantation as part of this clinical trial.
Arm/Group | Hematopoietic Stem Cell Transplantation
Serious Adverse Events (participants affected / at risk) | 10/36
Other Adverse Events (participants affected / at risk) | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hematopoietic Stem Cell Transplantation (N=36)
Syncopal Episode (Nervous system disorders) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
cerebral venous thrombosis and hemorrhage (Vascular disorders) | 1 (1)
aortic valve endocarditis (Cardiac disorders) | 1 (1)
pulmonary/upper respiratory chest pain (General disorders) | 1 (1)
progressive non-oliguric renal failure (Renal and urinary disorders) | 1 (1)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
norovirus (Infections and infestations) | 1 (1)
thrombosis/embolism (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hematopoietic Stem Cell Transplantation (N=36)
abdominal cramping (Gastrointestinal disorders) | 12 (12)
abdominal discomfort/tenderness (Gastrointestinal disorders) | 9 (9)
abdominal distention (General disorders) | 2 (2)
abdominal pain (Gastrointestinal disorders) | 16 (16)
aggitation (Psychiatric disorders) | 2 (2)
Alkaline Phosphatase (Investigations) | 22 (22)
ALT (Hepatobiliary disorders) | 26 (26)
anal/rectal erythema (Skin and subcutaneous tissue disorders) | 2 (2)
ANC (Blood and lymphatic system disorders) | 29 (29)
anemia (Blood and lymphatic system disorders) | 27 (27)
ankle pain (Musculoskeletal and connective tissue disorders) | 7 (7)
anorexia (Metabolism and nutrition disorders) | 15 (15)
anxiety (Psychiatric disorders) | 25 (25)
AST (Hepatobiliary disorders) | 30 (30)
back pain (Musculoskeletal and connective tissue disorders) | 9 (9)
basilar crackles (Respiratory, thoracic and mediastinal disorders) | 2 (2)
BK virus (Renal and urinary disorders) | 6 (6)
bloody stool (Gastrointestinal disorders) | 2 (2)
blurry vision (Eye disorders) | 5 (5)
BPH (Reproductive system and breast disorders) | 2 (2)
bradycardi (Cardiac disorders) | 2 (2)
bruising (Skin and subcutaneous tissue disorders) | 10 (10)
C diff (Infections and infestations) | 4 (4)
chest pain (General disorders) | 7 (7)
chest tightness (General disorders) | 6 (6)
chills (Investigations) | 18 (18)
cholecystitis (Gastrointestinal disorders) | 2 (2)
citrobacteria infection (Infections and infestations) | 2 (2)
CMV (Infections and infestations) | 18 (18)
confusion (Psychiatric disorders) | 6 (6)
conjunctivitis (Eye disorders) | 2 (2)
constipation (Gastrointestinal disorders) | 15 (15)
cough (Respiratory, thoracic and mediastinal disorders) | 25 (25)
increased creatinine (Metabolism and nutrition disorders) | 29 (29)
CVC drainage (Skin and subcutaneous tissue disorders) | 2 (2)
CVC pain/tenderness (Skin and subcutaneous tissue disorders) | 6 (6)
deconditioned (Musculoskeletal and connective tissue disorders) | 3 (3)
decreased appetite (Metabolism and nutrition disorders) | 19 (19)
decreased oral intake (Metabolism and nutrition disorders) | 3 (3)
dehydration (Metabolism and nutrition disorders) | 6 (6)
depression (Psychiatric disorders) | 12 (12)
diaphoresis (Metabolism and nutrition disorders) | 2 (2)
diarrhea (Gastrointestinal disorders) | 34 (34)
difficulty swallowing (Gastrointestinal disorders) | 6 (6)
diminished breath sounds (Respiratory, thoracic and mediastinal disorders) | 5 (5)
disoriented (Psychiatric disorders) | 3 (3)
dizziness/lighheadedness (General disorders) | 17 (17)
drowsiness (General disorders) | 9 (9)
dry eyes (Eye disorders) | 7 (7)
dry heaves (Gastrointestinal disorders) | 2 (2)
dry mouth (Gastrointestinal disorders) | 8 (8)
dry skin (Skin and subcutaneous tissue disorders) | 11 (11)
DVT (Vascular disorders) | 2 (2)
dyspepsia (Gastrointestinal disorders) | 11 (11)
dyspenea on exertion (Respiratory, thoracic and mediastinal disorders) | 5 (5)
dysuria (Renal and urinary disorders) | 4 (4)
ear congestion (Ear and labyrinth disorders) | 3 (3)
ear pain (Ear and labyrinth disorders) | 3 (3)
eczema (Skin and subcutaneous tissue disorders) | 2 (2)
edema (Blood and lymphatic system disorders) | 9 (9)
epistaxis (General disorders) | 12 (12)
erythema (Skin and subcutaneous tissue disorders) | 5 (5)
erythema at CVC site (Skin and subcutaneous tissue disorders) | 2 (2)
esophagitis (Gastrointestinal disorders) | 2 (2)
facial drooping (General disorders) | 2 (2)
facial redness (Skin and subcutaneous tissue disorders) | 3 (3)
facial swelling (General disorders) | 3 (3)
fall (Injury, poisoning and procedural complications) | 2 (2)
fatigue (General disorders) | 31 (31)
feeling "cold" (General disorders) | 2 (2)
fever (General disorders) | 29 (29)
flank pain (General disorders) | 2 (2)
flat affect (Psychiatric disorders) | 4 (4)
fluid overload (Blood and lymphatic system disorders) | 2 (2)
fluid retention (Blood and lymphatic system disorders) | 2 (2)
FLUSHING (General disorders) | 2 (2)
FOLLICULITIS (Skin and subcutaneous tissue disorders) | 2 (2)
FUNGAL RASH (Skin and subcutaneous tissue disorders) | 3 (3)
gas pain (Gastrointestinal disorders) | 2 (2)
gastritis (Gastrointestinal disorders) | 2 (2)
GERD (Gastrointestinal disorders) | 17 (17)
GI distress (Gastrointestinal disorders) | 7 (7)
gout (Immune system disorders) | 3 (3)
gram positive bacteremia (Infections and infestations) | 2 (2)
hallucinations (Psychiatric disorders) | 2 (2)
hand foot syndrome (Infections and infestations) | 3 (3)
headache/migraine (General disorders) | 26 (26)
hematuria (Renal and urinary disorders) | 5 (5)
hemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
hemorrhoids (Gastrointestinal disorders) | 6 (6)
hip pain (Musculoskeletal and connective tissue disorders) | 2 (2)
hsv (Infections and infestations) | 3 (3)
hyperbilirubinemia (Hepatobiliary disorders) | 11 (11)
hypercalcemia (Metabolism and nutrition disorders) | 11 (11)
hyperglycemia (Metabolism and nutrition disorders) | 30 (30)
hyperkalemia (Metabolism and nutrition disorders) | 18 (18)
hypermagnesemia (Metabolism and nutrition disorders) | 7 (7)
hypernatremia (Metabolism and nutrition disorders) | 12 (12)
hyperphosphatemia (Metabolism and nutrition disorders) | 2 (2)
hypertension (Cardiac disorders) | 21 (21)
hypoalbuminemia (Metabolism and nutrition disorders) | 28 (28)
hypocalemia (Metabolism and nutrition disorders) | 25 (25)
hypoglycemia (Metabolism and nutrition disorders) | 3 (3)
hypokalemia (Metabolism and nutrition disorders) | 23 (23)
hypomagnesemia (Metabolism and nutrition disorders) | 30 (30)
hyponatremia (Metabolism and nutrition disorders) | 25 (25)
hypophosphatemia (Metabolism and nutrition disorders) | 3 (3)
hypotension (Cardiac disorders) | 15 (15)
hypothyroidism (Endocrine disorders) | 3 (3)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 8 (8)
incontinent (stool) (Gastrointestinal disorders) | 4 (4)
increased thirst (General disorders) | 2 (2)
insomnia (Psychiatric disorders) | 18 (18)
leg/knee pain (Musculoskeletal and connective tissue disorders) | 6 (6)
limited range of motion (Musculoskeletal and connective tissue disorders) | 2 (2)
lip sore (General disorders) | 2 (2)
loss of balance (General disorders) | 4 (4)
lower extremity edema (Blood and lymphatic system disorders) | 11 (11)
malaise (General disorders) | 4 (4)
memory changes (Nervous system disorders) | 2 (2)
mouth erythema (Gastrointestinal disorders) | 2 (2)
mouth pain/tenderness (Gastrointestinal disorders) | 5 (5)
MRSE (Infections and infestations) | 8 (8)
mucositis (Gastrointestinal disorders) | 21 (21)
muscle spasm (Musculoskeletal and connective tissue disorders) | 3 (3)
myalgia/arthralgia (Musculoskeletal and connective tissue disorders) | 9 (9)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 (6)
nausea (Gastrointestinal disorders) | 33 (33)
neck pain (Musculoskeletal and connective tissue disorders) | 4 (4)
neutropenic fever (General disorders) | 4 (4)
night sweats (Investigations) | 5 (5)
nocturia (Renal and urinary disorders) | 2 (2)
pain (General disorders) | 8 (8)
pale skin (Skin and subcutaneous tissue disorders) | 2 (2)
parainfluenza (Infections and infestations) | 6 (6)
periorbital edema (Eye disorders) | 3 (3)
peripheral neuropathy (Nervous system disorders) | 11 (11)
PICC line erythema (Skin and subcutaneous tissue disorders) | 2 (2)
platelet reaction (Blood and lymphatic system disorders) | 2 (2)
pneumonia (Infections and infestations) | 5 (5)
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
post nasal drip (Respiratory, thoracic and mediastinal disorders) | 6 (6)
pruritis (Skin and subcutaneous tissue disorders) | 26 (26)
PTT (Blood and lymphatic system disorders) | 2 (2)
pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2 (2)
pulmonary nodules (Respiratory, thoracic and mediastinal disorders) | 3 (3)
rash (Skin and subcutaneous tissue disorders) | 26 (26)
rectal bleeding (Gastrointestinal disorders) | 3 (3)
rectal pain/discomfort (Gastrointestinal disorders) | 4 (4)
renal failure (Renal and urinary disorders) | 2 (2)
renal insufficiency (Renal and urinary disorders) | 9 (9)
respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4)
rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 8 (8)
rigors (General disorders) | 5 (5)
scratchy throat (General disorders) | 2 (2)
seasonal allergies (Respiratory, thoracic and mediastinal disorders) | 9 (9)
shaky (General disorders) | 2 (2)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 6 (6)
shoulder discomfort/pain (Musculoskeletal and connective tissue disorders) | 7 (7)
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 9 (9)
sinus drainage (Respiratory, thoracic and mediastinal disorders) | 5 (5)
sinus pressure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
sinus thickening (Respiratory, thoracic and mediastinal disorders) | 2 (2)
sinusitis (Respiratory, thoracic and mediastinal disorders) | 7 (7)
skin abrasion (Skin and subcutaneous tissue disorders) | 2 (2)
skin erythema (Skin and subcutaneous tissue disorders) | 2 (2)
skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
skin wound (Skin and subcutaneous tissue disorders) | 2 (2)
shortness of breath with exertion (Skin and subcutaneous tissue disorders) | 3 (3)
somnolence (General disorders) | 3 (3)
sore throat (Gastrointestinal disorders) | 15 (15)
staph bacteremia (Infections and infestations) | 2 (2)
steroid induced diabetes (Endocrine disorders) | 4 (4)
steroid myopathy (Musculoskeletal and connective tissue disorders) | 2 (2)
swelling at CVC (Skin and subcutaneous tissue disorders) | 2 (2)
swelling of the neck (General disorders) | 2 (2)
swelling of upper extremities (General disorders) | 2 (2)
syncope (General disorders) | 3 (3)
tachycardia (Cardiac disorders) | 17 (17)
taste alterations (Gastrointestinal disorders) | 9 (9)
thrombocytopenia (Blood and lymphatic system disorders) | 31 (31)
tonsillar adenopathy (Gastrointestinal disorders) | 2 (2)
tremors (General disorders) | 10 (10)
unsteady gait/balance (General disorders) | 3 (3)
upper extremity weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
URI (Respiratory, thoracic and mediastinal disorders) | 2 (2)
urinary frequency (Renal and urinary disorders) | 10 (10)
urinary hesitancy (Renal and urinary disorders) | 3 (3)
urinary incontinence (Renal and urinary disorders) | 5 (5)
urinary retention (Renal and urinary disorders) | 2 (2)
urinary urgency (Renal and urinary disorders) | 5 (5)
visual changes (Eye disorders) | 3 (3)
vomitting (Gastrointestinal disorders) | 27 (27)
VRE (Infections and infestations) | 3 (3)
watery eyes (Eye disorders) | 2 (2)
WBC (Blood and lymphatic system disorders) | 31 (31)
weakness (Musculoskeletal and connective tissue disorders) | 19 (19)
weight loss (Metabolism and nutrition disorders) | 7 (7)
wheezing (Respiratory, thoracic and mediastinal disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No